CLINICAL TRIAL: NCT02396719
Title: A Prospective, Single-Arm, Multicenter, Registry Study to Investigate the Performance of Femtosecond Laser-Assisted Cataract Surgery in Chinese Cataract Patients
Brief Title: A Real-World Registry to Investigate the Performance of LenSx® Laser in Chinese Patients
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CTO130-P001
Record Dates: First submitted 2015-03-19; First posted 2015-03-24 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LenSx: Phacoemulsification cataract surgery in at least 1 eye using LenSx® Laser technology
  Interventions: Device: LenSx® Laser

INTERVENTIONS:
Device: LenSx® Laser — Used for cornea incision, capsulotomy and lens fragmentation during cataract surgery

SUMMARY:
The purpose of this study is to investigate the performance of LenSx® Laser in femtosecond laser-assisted cataract surgery (FLACS) in real-world medical practice in Chinese patients.

DETAILED DESCRIPTION:
All subjects will undergo FLACS using the LenSx® Laser system. The recommended postoperative visits will follow the current standard of care in China.

ELIGIBILITY:
Inclusion Criteria:

* Chinese;
* Will undergo LenSx® Laser-assisted cataract surgery and phacoemulsification in at least one eye;
* Must sign written informed consent;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Contraindications listed in LenSx® Laser System Operator's Manual;
* Pregnant, nursing, or planning a pregnancy;
* Concurrent enrollment in another investigational drug and/or device study or participation in such a study within 30 days prior to surgery day;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients who undergo cataract surgery using LenSx® Laser and phacoemulsification in at least one eye will be eligible to participate.
Sampling Method: Probability Sample
Enrollment: 1541 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Completion rate of a round anterior capsulotomy | Surgery (Day 0)

SECONDARY OUTCOMES:
Completion rate of lens fragmentation without additional segmentation after LenSx Laser procedure | Surgery (Day 0)
Completion rate of intraocular lens (IOL) implantation | Surgery (Day 0)
Completion rate of corneal incisions | Surgery (Day 0)
Best-corrected distance visual acuity (BCDVA) | Up to Day 30
Percentage of patients with BCDVA of 20/20, 20/25, 20/40 or better at each visit | Up to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Zuojun Gao, Medical Affairs Director, Study Director — Alcon China
Locations (1):
- Alcon China Ophthalmic Product Co., Ltd., Beijing, China